CLINICAL TRIAL: NCT01057017
Title: Panitumumab and Bevacizumab Maintenance After First-Line FOLFOX-Bevacizumab for Patients With Advanced Colorectal Cancer With Wild-Type Ras
Brief Title: First-Line FOLFOX-Bevacizumab for Advanced Colorectal Cancer With Wild-Type Ras
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: possible lack of efficacy
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, howard safran, Director of BrUOG, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-CR-218
Record Dates: First submitted 2010-01-20; First posted 2010-01-27 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Methods; Bevacizumab; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): Bevacizumab: 7.5mg/kg, IV over 30-90 minutes every 3 weeks until disease progression.
  Panitumumab Dose Level 1: 6mg/kg over 60-120 minutes every 3 weeks until disease progression Dose Level 2: 9mg/kg over 60-120 minutes every 3 weeks until disease progression
  Interventions: Biological: intervention

INTERVENTIONS:
Biological: intervention
  Other Names: Bevacizumab: 7.5mg/kg, IV over 30-90 minutes every 3 weeks until disease progression.; Panitumumab; Dose Level 1: 6mg/kg over 60-120 minutes every 3 weeks until disease progression; Dose Level 2: 9mg/kg over 60-120 minutes every 3 weeks until disease progression

SUMMARY:
Bevacizumab given at 7.5mg/kg. IV over 10-90 minutes every 3 weeks until disease progression.Panitumumab given at 9mg/kg. IV over 30-90 minutes every 3 weeks until disease progression.Primary Objective: To determine the safety of every 3 week panitumumab and bevacizumab as maintenance therapy for patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
26 patients with advanced colorectal cancer will be given Bevacizumab at 7.5mg/kg. IV over 10-90 minutes every 3 weeks until disease progression.Panitumumab given at 9mg/kg. IV over 30-90 minutes every 3 weeks until disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or pathologically confirmed advanced colorectal cancer who received FOLFOX/bevacizumab for first-line treatment of metastatic disease.
2. Patients must not have had disease progression while receiving a minimum of 6 treatments of FOLFOX/bevacizumab. Patients with stable or responding disease on FOLFOX/bevacizumab are eligible. Bevacizumab does not need to be administered with all cycles of FOLFOX.
3. At least 3 weeks since prior FOLFOX/bevacizumab.
4. Wild type ras
5. No potentially curative treatment option.
6. ECOG performance status 0-1
7. Age>18, not pregnant or breast-feeding
8. Required entry laboratory parameters within 14 days of study entry: Granulocytes ≥ 1500/µl; platelet count ≥ 100,000/µl, Creatinine ≤ 2.0 mg/dl, Bilirubin ≤ 1.5 x upper limit of normal, AST ≤ 3 x upper limit of normal (or ≤ 5 x upper limit of normal for patients with liver metastases), Magnesium > lower limit of normal
9. Life expectancy of at least 16 weeks
10. Must not have uncontrolled severe, intercurrent illness.
11. No chemotherapy or radiation therapy within last 3 weeks
12. No concurrent anticancer therapy.
13. Signed study-specific consent form prior to study entry

Exclusion Criteria:

1. Prior EGFR inhibitor and prior irinotecan.
2. Clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >150/90 mmHg on medication], history of myocardial infarction within 6 months,), New York Heart Association (NYHA) Class II or greater congestive heart failure within 6 months, unstable arrhythmia. Patients with an atrial arrhythmia must have this condition well controlled on stable medication. Patients with current or recent (within 6 months) unstable angina are also not eligible.
3. Significant bleeding diathesis or coagulopathy
4. Major surgical procedure within 28 days prior to start of treatment. Port-a-cath placements are allowed.
5. Serious, nonhealing wound, ulcer, or current healing fracture
6. History of cerebral aneurysms or cerebral arteriovenous malformations.
7. Patients with recent (within 12 months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), or clinically significant peripheral artery disease should also be excluded.
8. Brain metastases
9. Patients with a history of a gastrointestinal fistula or perforation.
10. Significant infection or other coexistent medical condition that would preclude protocol therapy.
11. Interstitial lung disease
12. Patients who have had an organ transplant
13. Known positive test(s) for HIV infection, hepatitis C virus, acute or chronic active hepatitis B infection
14. Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
15. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, bladder and cervix are permissible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: howard p safran, MD, Principal Investigator — lifespan Hospitals
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 Patients were enrolled at The Miriam and Rhode Island Hospital
Groups:
- Panitumumab and Bevacizumab: Bevacizumab: 7.5mg/kg, IV over 30-90 minutes every 3 weeks until disease progression.
  Panitumumab Dose Level 1: 6mg/kg over 60-120 minutes every 3 weeks until disease progression Dose Level 2: 9mg/kg over 60-120 minutes every 3 weeks until disease progression
Period: Overall Study
Arm/Group | Panitumumab and Bevacizumab
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Toxicity to Combination of Panitumumab and Bevacizumab
Description: To determine the safety of every 3 week panitumumab and bevacizumab as maintenance therapy for patients with metastatic colorectal cancer. Use of CTCAE version 3
Time Frame: every 3 weeks until patient comes off study (progressive disease), for up to 2 years
Measure: Number; unit: participants
Arm/Group | Panitumumab and Bevacizumab
Number analyzed (Participants) | 5
participants | 1

ADVERSE EVENTS:
Time Frame: from time of signing consent to 30 days post last dose of drug (occurred up to approximately 10 months)
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5)
Anorexia (3), nausea(3), vomiting(2), weakness(3), confusion(1), hypok(3), hypophos(3), hypoca(3) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=5)
Fatigue (Investigations) | 2 (2)
Rash (Investigations) | 4 (4)
Skin Redness (Investigations) | 1 (1)
Constipation (Investigations) | 1 (1)
Yeast Infection (Investigations) | 1 (1)
Alk Phos (Investigations) | 1 (1)
AST (Investigations) | 1 (1)
dehydration (Investigations) | 1 (1)
abd pain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No